CLINICAL TRIAL: NCT01921322
Title: Sensor Augmented Pump Therapy Versus Multiple Daily Injection Therapy for Hospitalized Patients in China With Type 2 Diabetes; Time to Target
Brief Title: Sensor Augmented Pump Therapy Versus Multiple Daily Injection Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP270
Record Dates: First submitted 2013-08-09; First posted 2013-08-13 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Subjects randomly assigned to undergo treatment using either the Paradigm 722 insulin pump or multiple daily insulin injections.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pump (Experimental): Paradigm 722 insulin pump used for insulin infusion and continuous glucose monitoring
  Interventions: Device: Pump
- MDI (Active Comparator): Multiple daily insulin injections used for treatment
  Interventions: Other: CGMS Gold

INTERVENTIONS:
Device: Pump — 722 Paradigm Real-Time System
  Arms: Pump
Other: CGMS Gold — Device used to collect retrospective sensor data, blinded to the subjects, to compare to the treatment arm
  Arms: MDI

SUMMARY:
This is a prospective, randomized (open label), multi-center and post-market study. The study is to compare effectiveness of sensor-augmented pump (SAP) therapy versus multiple daily injection (MDI) therapy in hospitalized patients with insulin treating type 2 diabetes in China

DETAILED DESCRIPTION:
Primary objective:

To compare the length of time to achieve target glucose range using Self-Monitoring Blood Glucose (SMBG), as reference method, with the 722 Paradigm Real-Time insulin pump versus MDI

Secondary Objectives:

To compare glycemic variability (using CGM as reference method) with the 722 Paradigm Real-Time insulin pump versus MDI

This is a prospective, randomized (open label), multi-center study. The clinical study staff will conduct screening tests according to inclusion/exclusion criteria in order to verify the subject's eligibility for the study.

Inpatient Period A patient is admitted into hospital for treatment of diabetes

Randomization

Subjects are randomized (at a 1:1 ratio) to group A or B in the study database. A total of 80 subjects will be randomized into 2 study groups:

* Group A will wear 722 Paradigm Real-Time System (treated with 24h per day insulin infusion)
* Group B will be on MDI and wear the CGMS-Gold (treated with 4 insulin injections).

It is anticipated that the total duration for the study will be within one year from site initiation to finalization of all data entry and monitoring.

Each subject will participate in the study approximately 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 to 65 years old at time of screening
2. A clinical diagnosis of type 2 diabetes > 6 months prior to the screening as determined by the Investigator,
3. Treating with insulin at least one injection per day prior to participate in the study
4. Glycosylated hemoglobin (A1C) > 8% at screening
5. Subject needs to be hospitalized to receive treatment for glucose management according to Endocrinologists' discretion
6. Subject is willing to follow protocol and underdo all study procedures
7. Subject is willing and able to provide informed written consent personally or by legal proxy

Exclusion Criteria:

1. Subject has known hypersensitivity to insulin or insulin infusion set
2. Subject has been treated with drugs with a known effect on BG within 8 weeks before enrollment other than diabetes medications such as insulin or oral agents.
3. random blood glucose is above 33 mmol/L
4. Subject is currently using real time CGM therapy prior to screening
5. Subject is currently using insulin pump therapy prior to screening
6. Female subject who is pregnant, or plans to become pregnant during the course of the study
7. Patients who are critically ill that must go to intensive critical care unit per Investigator discretion
8. Subject has any systemic disease or medical condition found on the screening tests that may interfere with the safety of the patient and efficacy of the study treatment, in the opinion of the Investigator, may preclude him/her from participating in the study. The following includes, but not limited to, those conditions:

   * Female subject has a positive serum pregnancy screening test
   * Subject has visually impaired or disability limits the use of RT-CGM.
   * Subject has any unresolved adverse skin condition in the area of sensor placement or device replacement (e.g., psoriasis, rash, Staphylococcus infection)
   * Subject has disease with a known effect on BG such as Active Graves' disease
   * Subject has a history of alcohol abuse
9. Any other condition, which may not be suitable for the study at physician's discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Chinese PLA General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Multiple Daily Injections: Multiple daily insulin injections used for treatment
Period: Overall Study
Arm/Group | Pump | Multiple Daily Injections
Started | 57 | 61
Completed | 42 | 44
Not Completed | 15 | 17

BASELINE CHARACTERISTICS:
Population: Amoung the study completers, four met the target range on or before the first day and one subjects blinded CGM data was lost due to removal of the devices battery. The five subjects were excluded from the final analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pump | Multiple Daily Injections | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (10.2) | 49 (9.6) | 50 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 25 | 24 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 40 | 41 | 81
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height (cm) [Mean (Standard Deviation); unit: cm] | 167 (8.1) | 168 (7.6) | 167 (7.8)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 71 (11.9) | 72 (10.7) | 71 (11.2)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 25 (3.1) | 25 (3.3) | 25 (3.1)
A1C (%) [Mean (Standard Deviation); unit: %] | 10 (1.6) | 10 (1.2) | 10 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Time to Target
Description: length of time to achieve target glucose range using Self-Monitoring Blood Glucose (SMBG), as reference method, with the 722 Paradigm Real-Time insulin pump versus Multiple Daily Injection
Time Frame: Up to 14 days in hospital
Population: subjects included in final analysis
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pump | Multiple Daily Injections
Number analyzed (Participants) | 40 | 41
days | 3.7 (1.1) | 6.3 (3.1)

2. Secondary Outcome: Glycemic Variability
Description: Glycemic variability (mean amplitude glycemic excursion) using CGM as reference method
Time Frame: Up to 14 days in hospital
Population: subjects incluced in final analysis
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pump | Multiple Daily Injections
Number analyzed (Participants) | 40 | 41
mmol/L | 3.55 (1.89) | 3.44 (1.85)

ADVERSE EVENTS:
Time Frame: up to 14 days in hospital
Arm/Group | Pump | Multiple Daily Injections
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/61
Other Adverse Events (participants affected / at risk) | 1/57 | 1/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pump (N=57) | Multiple Daily Injections (N=61)
bleeding (General disorders) | 1 (1) | 0 (0)
allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No